CLINICAL TRIAL: NCT04201912
Title: Role of TLR2 and TLR4 in Stage 2 Periodontitis Patients With and Without Type 2 Diabetes
Brief Title: Role of TLR2 and TLR4 in Stage 2 Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Assistant Professor, Ajman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: D-F-19-03-03
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Periodontal Inflammation

STUDY DESIGN:
Intervention Model Description: Selection of patients by grading the patients according to criteria patients without periodontal and systemic involvement(control), patients classified as stage 2 periodontitis without systemic involvement(test group1), patients classified as stage 2 Periodontitis with systemic disease(Type 2 diabetes)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control patients (Placebo Comparator): Evaluation of Toll like receptor activity from whole saliva obtained from control patients
  Interventions: Diagnostic Test: saliva analysis for Toll like receptor activity
- Periodontal patients without diabetes (Active Comparator): Evaluation of toll like receptor activity from whole saliva obtained from periodontal patients without diabetes
  Interventions: Diagnostic Test: saliva analysis for Toll like receptor activity
- Periodontal patients with diabetes (Active Comparator): Evaluation of toll like receptor activity from whole saliva obtained from periodontal patients with diabetes
  Interventions: Diagnostic Test: saliva analysis for Toll like receptor activity

INTERVENTIONS:
Diagnostic Test: saliva analysis for Toll like receptor activity — Stimulated whole saliva will be obtained from patients and tested for Toll like receptor activity

SUMMARY:
In Health, mucosal inflammation is prevented by TLR (Toll like receptors) that interact with Specific MAMP (microbe associated molecular pattern). Currently about 13TLRs have been identified. Among them, TLR2 and 4 recognize most organisms . Periodontal disease is mixed infection resulting due to dysbiosis . When aggravated by systemic disease the role of TLRs is detrimental for the overall state of periodontal apparatus. Type 2 diabetes is one of the systemic disease which is seen a risk factor if uncontrolled can exaggerate the titer of TLR2 and TLR4 biomarkers . Various studies have been evaluated to determine the role of TLRs in autoimmune and periodontal conditions. The purpose of this study is to determine if both TLR2 and TLR4 play equal roles in periodontal disease and in cases where periodontal disease is complicated by the presence of systemic disease. Individual role of TLR2 and TLR4 in active disease will help determine treatment strategies and will also be able to predict potential biomarker in disease.

DETAILED DESCRIPTION:
In Health, mucosal inflammation is prevented by TLR (Toll like receptors) that interact with Specific MAMP (microbe associated molecular pattern). Currently about 13TLRs have been identified. Among them, TLR2 and 4 recognize most organisms. Periodontal disease is mixed infection resulting due to dysbiosis. When aggravated by systemic disease the role of TLRs is detrimental for the overall state of periodontal apparatus. Type 2 diabetes is one of the systemic disease which is seen a risk factor if uncontrolled can exaggerate the titer of TLR2 and TLR4 biomarkers. Various studies have been evaluated to determine the role of TLRs in autoimmune and periodontal conditions. The purpose of this study is to determine if both TLR2 and TLR4 play equal roles in periodontal disease and in cases where periodontal disease is complicated by the presence of systemic disease. Individual role of TLR2 and TLR4 in active disease will help determine treatment strategies and will also be able to predict potential biomarker in disease.

Periodontal diseases are classified according to the American academy of periodontology as stage 1, 2, 3&4 according to severity and extent of the disease progression.

Stage 2 periodontitis was selected as it is considered as an intermediary, because CAL(clinical attachment loss was standardized at 3-4mm,this could reflect the progression of disease and its impact from a horizontal bone loss to a more oblique one, if in case the dysbiosis persists.

ELIGIBILITY:
Inclusion Criteria:

* *Untreated stage 2 periodontitis patients (n-60)-Age group 21-60

  * Non Smokers
  * Diabetic patients controlled
  * Not haven taken medications in the past 3 months

Exclusion Criteria:

* smoker

  * habits such as betel, tobacco chewing
  * systemically unstable, Diabetes uncontrolled patients
  * haven taken medications in the past 3 months
  * Pregnant ladies
  * Periodontal involvement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Toll like receptor 2 activity | From baseline to 5 months
  Toll like receptor 2 activity will be measured from saliva obtained from controls, patients with periodontal disease but no diabetes and periodontal patients with diabetes

SECONDARY OUTCOMES:
Toll like receptor 4 activity | From baseline to 5 months
  Toll like receptor 4 activity will be measured from saliva obtained from controls, patients with periodontal disease but no diabetes and periodontal patients with diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Ajman University, Ajman, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided